CLINICAL TRIAL: NCT04904835
Title: Evaluation of the Beckman Coulter Access Hepatitis B Virus (HBV) Serological Marker Assays As an Aid in the Diagnosis of HBV Infection: EU Clinical Trial Protocol
Brief Title: Access HBV Assays - European Union (EU) Clinical Trial Protocol -
Status: Recruiting | Type: Observational
Sponsor: Beckman Coulter, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DC-TR18-0408; HBV-EU-08-19 (Other: Beckman Coulter, Inc)
Record Dates: First submitted 2021-05-18; First posted 2021-05-27 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: HBV
Keywords: Hepatitis B surface Antigen (HBsAg); Total hepatitis B core Antibody (HBcT); Hepatitis B e Antigen (HBeAg); Hepatitis B e Antibody (HBeAb); Hepatitis B surface Antibody (HBsAb); IgM Antibody to hepatitis B core Antigen (HBc IgM)
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (10):
- Unselected blood donors: leftover samples from unselected blood donors from at least 2 donation centers. Leftover samples to be tested by Access HBV serological marker assays and CE-marked (european compliance marked) predicate assays
  Interventions: Diagnostic Test: Access HBV serological marker assays on the DxI 9000 Access Immunoassay Analyzer and CE-marked predicate assays
- Hospitalized patients: Leftover samples to be tested by Access HBV serological marker assays and CE-marked predicate assays
  Interventions: Diagnostic Test: Access HBV serological marker assays on the DxI 9000 Access Immunoassay Analyzer and CE-marked predicate assays
- Presumed HBsAg positive patients: Leftover samples from patients at different stages of HBV infection (acute and chronic, minimum 10 per stage of infection), HBsAg positive by a Confirmatory testing of a CE-marked assay, including ≥ 25 "same day" fresh samples (tested ≤1 day after sampling), and minimum 20 high positive samples (>26 IU/mL) and minimum 20 samples in the cut-off range. If not enough samples in the cut-off range are obtained during the clinical trial, additional HBsAg specimens in the cut-off range will be tested by Research &Development to fit with Common Technical Specification requirements.
  Leftover samples to be tested by Access HBsAg assays and CE-marked predicate assays
  Interventions: Diagnostic Test: Access HBV serological marker assays on the DxI 9000 Access Immunoassay Analyzer and CE-marked predicate assays
- Patients having recovered from natural HBV infection, presumed Anti-HBs positive: Leftover samples from Patients positive for Anti-HBs and Anti-HBc Total by CE-marked assays. Target is to have at least ¾ of them recovered without HBV antiviral treatment.
  Leftover samples to be tested by Access anti-HBs assay and CE-marked predicate assays
  Interventions: Diagnostic Test: Access HBV serological marker assays on the DxI 9000 Access Immunoassay Analyzer and CE-marked predicate assays
- Patients having received HBV vaccination, presumed Anti-HBs positive: Leftover samples Confirmed as vaccinated by testing at the time of enrollment (i.e. positive for Anti-HBs and negative for Anti-HBc by CE-marked assays).Leftover samples to be tested by Access anti-HBs assay and CE-marked predicate assays
  Interventions: Diagnostic Test: Access HBV serological marker assays on the DxI 9000 Access Immunoassay Analyzer and CE-marked predicate assays
- Presumed Anti-HBc Total positive patients: Leftover samples from Patients at different stage of infection (acute, chronic or recovered, minimum 10 per stage of infection) positive for Anti-HBc Total by a CE-marked assay, including ≥ 25 "same day" fresh samples (tested ≤1 day after sampling).
  Leftover samples to be tested by Access anti-HBc Total and CE-marked predicate assays
  Interventions: Diagnostic Test: Access HBV serological marker assays on the DxI 9000 Access Immunoassay Analyzer and CE-marked predicate assays
- Presumed Anti-HBc IgM positive patients: left over samples from Patients with acute/recent HBV infection, positive for Anti-HBc IgM by a CE-marked assay.
  Leftover samples to be tested by Access anti-HBc IgM assay and CE-marked predicate assays
  Interventions: Diagnostic Test: Access HBV serological marker assays on the DxI 9000 Access Immunoassay Analyzer and CE-marked predicate assays
- Presumed HBeAg positive patients: Leftover samples from Patients at different stages of infection (acute and chronic, minimum 5 per stage of infection), positive for HBeAg by a CE-marked assay.
  Leftover samples to be tested by Access HBeAg assay and CE-marked predicate assays
  Interventions: Diagnostic Test: Access HBV serological marker assays on the DxI 9000 Access Immunoassay Analyzer and CE-marked predicate assays
- Presumed Anti-HBe positive patients7: Leftover samples from Patients at different stages of infection (chronic and recovered, minimum 5 per stage of infection), positive for Anti-HBe by a CE-marked assay.
  Leftover samples to be tested by Access anti-HBe assay and CE-marked predicate assays
  Interventions: Diagnostic Test: Access HBV serological marker assays on the DxI 9000 Access Immunoassay Analyzer and CE-marked predicate assays
- Patients with chronic HBV infection: Leftover samples to be tested by Access anti-HBc IgM assay and CE-marked predicate assay
  Interventions: Diagnostic Test: Access HBV serological marker assays on the DxI 9000 Access Immunoassay Analyzer and CE-marked predicate assays

INTERVENTIONS:
Diagnostic Test: Access HBV serological marker assays on the DxI 9000 Access Immunoassay Analyzer and CE-marked predicate assays — All samples will be tested with both CE-marked HBV serological predicate assays (HBsAg, HBsAb, HBcT, HBc IgM, HBeAb, and/or HBeAg assays) and Access HBV serological assays (HBsAg, HBsAb, HBcT, HBc IgM, HBeAb, and/or HBeAg assays) according to respective Instructions For Use to determine non-reactive (NR), initially reactive (IR), repeatedly reactive (RR), or confirmed or not confirmed Positive.

SUMMARY:
The objective of this protocol is the collection and testing of clinical samples to determine the clinical performance of the Access HBV serological marker assays on the DxI 9000 Access Immunoassay Analyzer.

The study will involve a multicenter, prospective and retrospective collection of samples, and testing of samples with the investigational Hepatitis B Virus assays as required per the European Union Common Technical Specification. All samples collected will be anonymized or pseudo-anonymised, leftover, remnant samples. Pseudo-anonymised collection of samples will require documented patient consent (oral or written).

DETAILED DESCRIPTION:
Sensitivity to final status on presumed HBV serological marker positive subjects will be calculated. Specificity will be calculated from hospitalized patients and blood donors specimens. False Initial Reactive Rate will be calculated on fresh hospitalized patient samples for Access HBsAg assay only (Qualitative).

ELIGIBILITY:
Inclusion Criteria:

* Subject aged ≥ 18 years,
* Subject who has provided consent (oral or written) or sample collected under waiver
* With sufficient volume to perform clinical trial testing
* And belonging to one of the following enrollment groups:

  * Unselected blood donors
  * Hospitalized patients
  * Presumed HBsAg positive patients by Confirmatory testing of a CE-marked assay
  * Patients having recovered from natural HBV infection, presumed Anti-HBs positive (i.e. Anti-HBs and Anti-HBc Total positive by CE-marked assays)
  * Patients having received HBV vaccination, presumed Anti-HBs positive (confirmed by testing at the time of enrollment, i.e. positive for Anti-HBs and negative for Anti-HBc by CE-marked assays).
  * Presumed Anti-HBc Total positive patients by a CE-marked assay
  * Presumed Anti-HBc IgM positive patients by a CE-marked assay with acute/recent HBV infection 8
  * Presumed HBeAg positive patients by a CE-marked assay
  * Presumed Anti-HBe positive patients by a CE-marked assay
  * Patients with chronic HBV infection

Exclusion Criteria:

* Samples from subjects already included in the study* (* Patient can be included only once per HBV marker study, but can potentially be enrolled for several separate HBV marker studies.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The test population includes :
  1. 16,400 Unselected blood donors from at least 2 donation centers
  2. 2,700 Hospitalized patients
  3. 450 Presumed HBsAg positive patients
  4. 150 Patients having recovered from natural HBV infection, presumed Anti-HBs positive
  5. 300 Patients having received HBV vaccination, presumed Anti-HBs positive
  6. 450 Presumed Anti-HBc Total positive patients
  7. 220 Presumed Anti-HBc IgM positive patients 8-220 Presumed HBeAg positive patients
  9- 220 Presumed Anti-HBe positive patients 10- 100 Patients with chronic HBV infection TOTAL n=21,210
Sampling Method: Non-Probability Sample
Enrollment: 21210 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy measured as sensitivity and specificity | Baseline
  The endpoint will be diagnostic accuracy measured as sensitivity and specificity of Access HBV serological assays compared to sample status determined by specific testing algorithm for each HBV marker

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Centre de Ressources Biologiques Biobanque de Picardie CHU Amiens-Picardie, Amiens
  - Etablissement Français du Sang (EFS) Hauts-de-France - Normandie, Bois-Guillaume
  - Eurofins Biomnis, Ivry-sur-Seine
  - Laboratoire de Virologie, Laboratoire associé au CNR du VIH Institut de Biologie Clinique ; hôpital C : Nicolle, CHU Rouen, Rouen
  - Cerba Xpert, Saint-Ouen-l'Aumône

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dzamitika S, Boulaire FL, Coignard C, Vincent C, Plantier JC, Lemee V, Greaume S, Voisin I, Brochot E, Herpe YE, Demirdjian G, Karagueuzian M, Afful D, Bayoud R, Hey J. Performance evaluation of the Access anti-HBc Total assay on the DxI 9000 Access Immunoassay Analyzer. Diagn Microbiol Infect Dis. 2024 Sep;110(1):116303. doi: 10.1016/j.diagmicrobio.2024.116303. Epub 2024 Apr 20. PMID 38838460